CLINICAL TRIAL: NCT04815993
Title: A Single Ascending Dose Trial to Assess the Pharmacokinetics, Safety, and Tolerability of Orally Administered SYN-020 Delayed Release Capsules in Healthy Subjects
Brief Title: Pharmacokinetics, Safety, and Tolerability of SYN-020
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theriva Biologics, Inc. (Industry)
Collaborators: Spaulding Clinical Research LLC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SB-1-020-001
Record Dates: First submitted 2021-03-12; First posted 2021-03-25 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Enteritis Caused by Radiation (Disorder)

STUDY DESIGN:
Intervention Model Description: single ascending dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SYN-020, 5 mg (Experimental): 6 subjects to receive a single 5 mg dose of SYN-020
  Interventions: Drug: SYN-020 delayed release capsule
- SYN-020, 15 mg (Experimental): 6 subjects to receive a single 15 mg dose of SYN-020
  Interventions: Drug: SYN-020 delayed release capsule
- SYN-020, 45 mg (Experimental): 6 subjects to receive a single 45 mg dose of SYN-020
  Interventions: Drug: SYN-020 delayed release capsule
- SYN-020, 150 mg (Experimental): 6 subjects to receive a single 150 mg dose of SYN-020
  Interventions: Drug: SYN-020 delayed release capsule

INTERVENTIONS:
Drug: SYN-020 delayed release capsule — SYN-020, is an opaque, white, size 3 HPMC capsule for oral administration containing enteric-coated, delayed-release pellets.
  Other Names: Intestinal Alkaline Phosphatase

SUMMARY:
This is a Phase 1, single-center, open-label, single ascending dose study to assess the PK, safety, and tolerability of SYN-020 delayed release capsules administered orally to healthy adult male and female subjects with a BMI of 18.5 to 27 kg/m2. Up to 36 subjects will participate, in each of up to 6 sequential cohorts. Single doses of 5, 15, 45, and 150 mg SYN-020 are planned in Cohorts 1 through 4, respectively. Cohorts 5 and 6, if enrolled, will receive doses that were well tolerated in an earlier cohort to determine the effect of BMI and/or a high-fat meal on the SYN-020 PK profile.

For each cohort, eligible subjects will be admitted to the clinic on Day -1, and receive study drug in the morning of Day 1. For PK analysis, blood and feces will be collected before dosing and for up to 96 hours (blood) or 120 hours (feces) after dosing. Subjects will be discharged from the clinic after the End of Study procedures are completed on Day 6.

DETAILED DESCRIPTION:
Intestinal alkaline phosphatase (IAP) is a naturally occurring enzyme produced by the small intestine in all mammals, including humans, and is considered essential for promoting normal gastrointestinal (GI) function and maintaining proper gut homeostasis, as well as appearing to play a pivotal role in the mediation of inflammation.

SYN-020 is a recombinant bovine IAP isotype II being developed by Synthetic Biologics, Inc. to reduce the cumulative GI toxicity and inflammation that can be associated with repeat administration of radiation in patients with cancer.

This is a Phase 1, single-center, open-label, single ascending dose study to assess the PK, safety, and tolerability of SYN-020 delayed release capsules administered orally to healthy adult male and female subjects with a BMI of 18.5 to 27 kg/m2. Up to 36 subjects will participate, with 6 subjects (approximately equal numbers of male and females) in each of up to 6 sequential cohorts. Single doses of 5, 15, 45, and 150 mg SYN-020 are planned in Cohorts 1 through 4, respectively. Cohorts 5 and 6, if enrolled, will receive doses that were well tolerated in an earlier cohort to determine the effect of BMI and/or a high-fat meal on the SYN-020 PK profile, and will be described fully in a protocol amendment.

For each cohort, eligible subjects will be admitted to the clinical research unit (CRU) on Day -1, and subjects who remain eligible will, after a minimum 10-hour overnight fast, receive study drug in the morning of Day 1. For PK analysis, blood and feces will be collected before dosing and for up to 96 hours (blood) or 120 hours (feces) after dosing. Subjects will be discharged from the CRU after the End of Study (EOS) procedures are completed on Day 6.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to read, write, and comprehend English at a sufficient level to understand study related materials, has provided written informed consent before any study-related procedure was performed, and is willing and able to comply with all testing and study requirements.
2. Subject is a healthy male or female, aged 18 through 50 years, inclusive.
3. Subject does not use any tobacco or nicotine product (eg, cigarette, pipe, e-cigarette, vape) and has not used any tobacco or nicotine product for at least 2 months before Day -1.
4. Subject has a BMI of 18.5 to 27 kg/m2 for initial cohorts or, for exploratory cohorts, ≥ 27.1 kg/m2. For Cohorts 1 through 4, if insufficient subjects are available to meet this criterion, subjects with a BMI up to 29 kg/m2 may be included with written authorization from the Sponsor.
5. Subject is healthy based on physical examination, clinical laboratory tests, 12-lead ECG, and vital signs.
6. Subject is willing to minimize the risk of inducing pregnancy from the time of signing the informed consent form (ICF) to at least either 90 days (males) or 30 days (females) after the study drug dose.
7. If female, subject has a negative serum pregnancy test at Screening and on Day -1 (CRU admission).
8. Subject usually has at least 1 bowel movement a day based on self-reporting.

Exclusion Criteria:

1. Subject has a history or the presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, vascular, metabolic, collagen, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
2. Subject has any known malabsorption syndrome or history of gastrointestinal surgery that could compromise the study objectives.
3. Subject has used any medication (prescription or non-prescription) or herbal supplement, other than prescription hormone replacement therapy (eg, thyroid, testosterone, estrogen) or contraception methods described in Inclusion Criterion #6, within 21 days before Day -1.
4. Subject is pregnant, breastfeeding, or not using a medically accepted method of contraception.
5. Subject is unable to abstain from artificial sweeteners (eg, aspartame, acesulfame potassium, advantame, saccharin, stevia, and sucralose) from CRU admission to the end of study participation.
6. Subject has a positive urine drug or alcohol test at Screening or CRU admission OR has a history of drug/alcohol abuse within 12 months before Screening.
7. Subject has donated more than 500 mL blood during the 3-month period before Day -1.
8. Subject has known intolerance of study drug/ingredients.
9. In the judgment of the Investigator, subject has any factor (eg, other treatment) that could invalidate the study result.
10. Subject is currently enrolled in another clinical study or has received an investigational drug or device within 30 days or within a time period consistent with a washout period of 5 half-lives before signing the ICF, whichever is longer.
11. Subject has already participated in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
SYN-020 systemic absorption | Daily Day 1 through Day 5
  Analysis of SYN-020 level present in blood
SYN-020 presence in feces | Daily Day -1 through Day 6
  Analysis of SYN-020 level present in feces

SECONDARY OUTCOMES:
Percentage of Participants with Changes in Clinical Laboratory Testing | Day -1, Day 2, Day 6
  Hematology, clinical chemistry, urinalysis, virus serology, drug screen, alcohol screen, pregnancy test, postmenopausal screen
Number of Participants With Changes in Physical exam | Day 1 and Day 6
  Complete and abbreviated physical examinations will be performed
Number of Participants with Changes in Vital Signs | Daily Day -1 through Day 6
  Blood pressure, pulse rate, respiratory rate, oral temperature
Number of Participants with Changes in Electrocardiograms | Day -1, Day 1, Day 2, Day 6
  12-lead ECG, P-wave, QRS-complex, QT-interval
Immunogenicity testing | Day 1, Day 6
  Measurement of anti-drug antibodies by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Sanabria, MD, Principal Investigator — Spaulding Clinical Research LLC
Locations (1):
- Spaulding Clinical Research LLC, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No